CLINICAL TRIAL: NCT04785989
Title: Metabolic Profiling of Leukemic Cells Through Isotope Tracing in Patients With CLL
Brief Title: In Vivo Metabolic Profiling of CLL (Chronic Lymphocytic Leukemia)
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: UW20062; MSN240796 (Other Grant/Funding Number: WISCONSIN ALUMNI RESEARCH FOUNDATION); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); A534260 (Other: UW Madison); Protocol Version 10/19/2022 (Other: UW Madison); 2020-1008 (Other: HSIRB UW Madison)
Record Dates: First submitted 2021-02-25; First posted 2021-03-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Cell metabolic tracing; Leukemic lymphocytes; Fuel preference
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Healthy volunteers: Healthy volunteers are defined as people without a history of cancer
  Interventions: Other: [U-13C]glucose
- Group B subset-1: Treatment naïve CLL(Chronic Lymphocytic Leukemia) patients with low disease burden: Participants with low disease burden CLL (Chronic Lymphocytic Leukemia) defined as confined to Rai stage 0.
  Interventions: Other: [13C5]glutamine
- Group B subset-2: Treatment naïve CLL patients with low disease burden: Participants with low disease burden CLL (Chronic Lymphocytic Leukemia) defined as confined to Rai stage 0.
  Interventions: Other: [U-13C]glucose
- Group C:Treatment naïve CLL patients with high systemic disease burden: Treatment naïve CLL patients with high systemic disease burden
  Interventions: Other: [U-13C]glucose

INTERVENTIONS:
Other: [U-13C]glucose — [U-13C]glucose will be administered as a bolus of 8 g (grams) over 10 minutes followed by 8 g/hour continuous infusion over 2 hours . This infusion rate will allow glucose tracer to reach sufficient enrichment without causing significant metabolic perturbation such as hyperglycemia.
  Groups: Group A: Healthy volunteers; Group B subset-2: Treatment naïve CLL patients with low disease burden; Group C:Treatment naïve CLL patients with high systemic disease burden
Other: [13C5]glutamine — 6mg/kg of body weight of [13C5]glutamine will be administered as a bolus over 10 minutes (± 1 minute) followed by 6mg/kg/hr body weight continuous infusion for 2 hours through a peripheral IV catheter/line. This infusion rate will allow glutamine tracer to reach sufficient enrichment without causing significant metabolic perturbation such as hyperglycemia.
  Groups: Group B subset-1: Treatment naïve CLL(Chronic Lymphocytic Leukemia) patients with low disease burden

SUMMARY:
Metabolic reprogramming has been identified as a hallmark of cancer. Almost a century after Otto Warburg initially discovered increased glycolytic activity in tumor tissue ("Warburg effect"), therapeutic targeting of cancer metabolism has become a field of intense research effort in cancer biology.

A growing appreciation of metabolic heterogeneity and complexity is currently reshaping investigators "simplistic" understanding of metabolic reprogramming in cancer. Discovering metabolic vulnerabilities as new treatment targets for cancer requires systematic dissection of metabolic dependencies, fuel preferences, and underlying mechanisms in the specific physiological context. However, today's data on cancer cell metabolic signatures and heterogeneity in their physiological habitat of the human organism is sparse to non-existent representing a critical knowledge gap in designing effective metabolic therapies. Here, the investigators propose a "top-down" approach studying cancer cell metabolism in patients followed by mechanistic in-depth studies in cell culture and animal models to define metabolic vulnerabilities.

Investigators will develop a metabolic tracing method to quantitatively characterize metabolic signatures and fuel preferences of leukemic lymphocytes in patients with chronic lymphocytic leukemia (CLL). Isotopic metabolic tracers are nutrients that are chemically identical to the native nutrient. Incorporated stable, non-radioactive isotopes allow investigators to follow their metabolic fate by monitoring conversion of tracer nutrients into downstream metabolites using cutting-edge metabolomics analysis. Using this method, investigators propose to test the hypothesis that leukemic lymphocytes show tissue-specific metabolic preferences that differ from non-leukemic lymphocytes and that ex vivo in-plasma labeling represents a useful model for assaying metabolic activity in leukemic cells in a patient-specific manner.

ELIGIBILITY:
Inclusion Criteria:

Group A

* Adult (18 years of age or older)
* No previous history of cancer
* Routine history of normal blood counts and vital signs
* Documented Informed Consent

Group B

* Adult (18 years of age or older)
* Diagnosis of CLL with low disease burden defined as Rai stage 0 ((Lymphocytosis; no enlargement of the lymph nodes, spleen, or liver; red blood cell and platelet counts are near normal.)
* Treatment naïve
* Documented Informed Consent

Group C

* Adult (18 years of age or older)
* Diagnosis of CLL with high systemic disease burden defined as infiltration of bone marrow causing cytopenia
* Treatment naïve
* Able/willing to have bone marrow aspiration
* Documented Informed Consent

Exclusion Criteria:

For all participants

* Prisoners
* Psychiatric inpatients or people who are institutionalized
* Minor (Less than 18 years of age)
* History of diabetes
* Cannot be on antihyperglycemic therapy
* Carbohydrate restricting diets: Atkins, Vegan, Ketogenic, etc.
* Females of child bearing potential
* Persons without decision-making capacity
* Person who cannot read/write English
* Not meeting inclusion criteria defined above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To meet the study aims sixteen (16) adult participants will be enrolled: four (4) healthy volunteers defined as people without a history of cancer, 8 patients with low disease burden CLL (Chronic Lymphocytic Leukemia) defined as confined to Rai stage 0, and 4 patients with high disease burden CLL defined as having extensive infiltration of the bone marrow.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Amount of [U-13C]glucose incorporation into metabolites in normal and leukemic lymphocytes: Liquid chromatography-mass spectrometry (LCMS) pharmacokinetic analysis | up to 2 hours (± 5 minutes)
  It will reveal how CLL cells utilize glucose compared to non-leukemic lymphocytes and how this changes with different disease burden and site of disease. Participants will be on overnight fasting.
Amount of [U-13C15N]L-glutamine incorporation into metabolites in normal and leukemic lymphocytes: LCMS pharmacokinetic analysis | up to 2 hours (± 5 minutes)
  It will reveal how CLL cells utilize glutamine compared to non-leukemic lymphocytes and how this changes with different disease burden and site of disease. Participants will be on overnight fasting.

OTHER OUTCOMES:
Validate ex vivo labeling model to assay metabolism | 10 minutes
  Study team seek to develop a more cost-effective ex vivo model to assay metabolism under conditions closest to the physiological setting in a small amount of blood. In addition, this model will allow numerous pharmacologic interventions and may serve as a personalized ex vivo drug screening assay.
  Participants will be on overnight fasting. Cells and plasma will be separated from 5 ml of pre infused blood. Cell suspensions will be incubated at 37°C for 2hrs and intracellular and extracellular metabolites will be extracted separately for LCMS analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Fletcher, MD, Principal Investigator — School of Medicine and Public Health, University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No